CLINICAL TRIAL: NCT01863485
Title: Phase 1 Safety, Tolerability, and Pharmacokinetic Study of CM082 (X-82) Tablets in Advanced Cancer Patients in China
Brief Title: Phase 1 Study of CM082 (X-82) Tablets in Advanced Cancer Patients in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AnewPharma (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM082-CA-I-001; 2013L00579、2013L00581 (Other: China FDA)
Record Dates: First submitted 2013-05-22; First posted 2013-05-29 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Advanced Cancer
Keywords: advanced cancer
MeSH Terms: interventions — vorolanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CM082 (Experimental): CM082 tablet
  Interventions: Drug: CM082 Tablet

INTERVENTIONS:
Drug: CM082 Tablet — CM082 tablets taken orally once a day on 28-day cycles
  Other Names: X-82

SUMMARY:
This is a Phase I Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CM082 tablets in Chinese Patients With Advanced Solid Tumors.

DETAILED DESCRIPTION:
This is a Phase I Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CM082 tablets in Chinese Patients With Advanced Solid Tumors. After the maximum tolerated dose (MTD) or the optimal biological dose is identified, an expansion cohort of ~20 advanced renal cell carcinoma patients will be enrolled to further characterize the safety and tumor response by CT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumor malignancy that is not responsive to standard therapies or for which there is no effective therapy.
* Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1.
* Life expectancy of at least 12 weeks.
* No immuno deficiency.
* Adequate organ system function, defined as follows:

  * Absolute neutrophil count (ANC) ≥1.5 x 10**9/L
  * Platelets ≥100 x 10**9/L
  * Hemoglobin ≥10 g/dL
  * Total bilirubin ≤1.5 times the upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5x the upper limit of normal (ULN) if no liver involvement or ≤2.5x the upper limit of normal with liver involvement.
  * Creatinine ≤ 1.5 x ULN.
* At least 4 weeks or 5 half-life after receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization.
* Willingness and ability to comply with trial and follow-up procedures.
* Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

* Not recovered from prior anti-cancer therapy or surgery.
* Have taken strong cytochrome P450 3A4 inhibitors or inducers in the last 2 weeks.
* Concomitant use of drugs with a risk of causing prolonged corrected QT interval and/or Torsades de Pointes.
* Patients with a history of intolerance to, or significant toxicity with, VEGFR tyrosine kinase inhibitor(s) (TKI).
* Females who are pregnant or breastfeeding.
* Those in reproductive ages who refuse to use contraception.
* Those with concurrent condition(e.g. psychological, neuronal, cardiovascular, respiratory conditions or infections) that in the investigator's opinion would jeopardize compliance with the protocol.
* Patients with known central nervous system (CNS) metastases.
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of CM082 (X-82).
* Patients with known GI disorders such as vomiting, diarrhea.
* Patients who are hepatitis B virus positive.
* Drug abuser.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months
  To determine the Maximum Tolerated Dose in Chinese patients with advanced solid tumors.

OTHER OUTCOMES:
Preliminary biological activity | 24 months
  clinical tumor response by computed tomography (CT) after treatment with CM082 tablets given as a single agent.
Area Under Curve | 2 months
Half-life time | 2 months
Cmax | 2 months
  Peak concentration
Tmax | 2 months
  Time to Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Wan Wang, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
Locations (3):
- China (3):
  - Beijing University First Hospital, Beijing, Beijing Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing